CLINICAL TRIAL: NCT06942767
Title: An Open-label, Multicenter Phase II Clinical Study of QLS31905 for Injection Combined With QL2107 Injection and XELOX Regimen in the First-line Treatment of CLDN18.2-positive Unresectable Locally Advanced or Metastatic Gastric or Gastroesophageal Junction (GEJ) Adenocarcinoma
Brief Title: Combination of QLS31905, QL2107 and Chemotherapy as First-line Therapy in CLDN18.2-positive Unresectable Locally Advanced or Metastatic Gastric or Gastroesophageal Junction (GEJ) Adenocarcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QLS31905-203
Record Dates: First submitted 2025-04-17; First posted 2025-04-24 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma
Keywords: CLDN18.2, gastric or gastroesophageal junction (GEJ) adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma | interventions — Injections; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QLS31905+QL2107+ XELOX (Experimental): QLS31905+QL2107+ oxaliplatin + capecitabine
  Interventions: Drug: QLS31905 for Injection; Drug: QL2107 Injection; Drug: Oxaliplatin Injection; Drug: Capecitabine Tablets

INTERVENTIONS:
Drug: QLS31905 for Injection — QLS31905 for Injection
Drug: QL2107 Injection — QL2107 Injection
Drug: Oxaliplatin Injection — Oxaliplatin Injection
Drug: Capecitabine Tablets — Capecitabine Tablets

SUMMARY:
This is an open-label, multicenter Phase II clinical study aimed at evaluating the tolerability, safety, efficacy, PK profile, and immunogenicity of QLS31905 for Injection combined with QL2107 Injection and XELOX regimen in the first-line treatment of CLDN18.2-positive unresectable locally advanced or metastatic gastric or gastroesophageal junction (GEJ) adenocarcinoma.

DETAILED DESCRIPTION:
QLS31905 is a bispecific antibody targeting CD3 and CLDN18.2 independently developed by Qilu Pharmaceutical Co., Ltd.

QL2107 is a biosimilar of pembrolizumab (Keytruda®) developed by Qilu Pharmaceutical Co., Ltd.

This is an open-label, multicenter Phase II clinical study aimed at evaluating the tolerability, safety, efficacy, PK profile, and immunogenicity of QLS31905 for Injection combined with QL2107 Injection and XELOX regimen in the first-line treatment of CLDN18.2-positive unresectable locally advanced or metastatic gastric or gastroesophageal junction (GEJ) adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with unresectable locally advanced or metastatic gastric or gastroesophageal junction (GEJ) adenocarcinoma confirmed by histopathological or cytological examination;
* Subjects with at least one measurable lesion designated as a target lesion, as assessed by the investigator according to RECIST v1.1. Lesions that have received radiotherapy or other local treatments may be considered measurable if they demonstrate imaging PD;
* No prior systemic anti-tumor treatment for locally advanced or metastatic gastric or gastroesophageal junction (GEJ) adenocarcinoma.

Exclusion Criteria:

* Subjects with a known history of severe or repeated allergy, intolerance, or contraindication to QLS31905, QL2107, or other large molecule protein preparations, as well as Oxaliplatin Injection or Capecitabine Tablets and any components in their preparations;
* Subjects had other second primary malignancies within 5 years prior to the first dose;
* Subjects with clinically significant hemorrhage within 3 months before the first dose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
DLT | up to 42 days following first dose
  Dose Limiting Toxicity，for Dose Escalation Stage
MTD | up to 42 days following first dose
  Maximum Tolerated Dose，for Dose Escalation Stage.
ORR (Objective Response Rate) | Approximately 24 months
  ORR is defined as the proportion of participants who have a best overall response of Complete Response (CR) or Partial Response (PR) as assessed by investigator per RECIST 1.1

SECONDARY OUTCOMES:
AE (adverse events) | Approximately 24 months
  AEs are any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of anti-drug antibody (ADA) Positive Participants | Approximately 24 months
  Immunogenicity will be measured by the number of participants that are ADA positive.
DOR (Duration of Response) | Approximately 24 months
  DOR is defined as the time from the date of the first response (CR/PR) until the date of radiological progressive disease or death due to any cause (whichever occurs first)
PFS (Progression Free Survival) | Approximately 24 months
  PFS is defined as the duration from the subject's first dose of the investigational product to the first imaging confirmation of radiological progressive disease or death due to any cause (whichever occurs first).
OS (Overall Survival) | Approximately 24 months
  OS is defined as the duration from the first dose of the investigational product to the time point when death occurs due to any cause.
Maximum concentration (Cmax) | Approximately 24 months
  Cmax will be derived from the PK serum samples collected.
Terminal elimination half-life (T1/2) | Approximately 24 months
  T1/2 will be derived from the PK serum samples collected.